CLINICAL TRIAL: NCT02516917
Title: The Feasibility of a Brief Attention Training Technique for Improving Behaviour and Attention in Children With ADHD
Brief Title: The Feasibility of a Brief Attention Training Technique in Improving Behaviour and Attention in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor of Clinical and Experimental Psychopathology, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 163562
Record Dates: First submitted 2015-07-31; First posted 2015-08-06 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

ARMS (1):
- Attention Training Technique (ATT) (Experimental): Participants will receive 3-5 sessions of the ATT over a period of 3-5 weeks. A set of standardised instructions will be read to each participant and then they will engage in the procedure for a period of 12 minutes. Participants will listen to a set of auditory stimuli and follow the directions of the recording. This will ask them to focus their attention on selected sounds or spatial locations, switch attention between different sounds and locations, before allocating their attention to all sounds simultaneously. Participants will be given a recording of the ATT on a C.D and asked to practice this at least once before the second session.
  Interventions: Behavioral: Attention Training Technique

INTERVENTIONS:
Behavioral: Attention Training Technique

SUMMARY:
This study aims to investigate the application of the Attention Training Technique in children with ADHD aged 7-11 years old. The research aims to investigate both the feasibility of this technique in this population as well as whether it can improve symptoms, behaviour and executive functioning.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is a neurobehavioural disorder characterised by core symptoms of hyperactivity, impulsivity and inattention. Its prevalence ranges between 3-9% of school-aged children, making it one of the most common presentations in child and adolescent mental health services.

In the last 10 years, research into the effectiveness of attention training as an intervention for children with ADHD has been increasing. This has tended to follow assumptions that children with the disorder either lack skills in focusing and maintaining their attention and/or have neurological deficits in areas responsible for attention functions. Results have been encouraging, with study participants demonstrating improvements in symptoms and behaviour following a course of attention training. However, the method and length of training has varied across studies.

This study aims to investigate a treatment called the Attention Training Technique (ATT) that approaches attention difficulties in this disorder from a different perspective. Instead of viewing inattention as a result of structural or skills deficits, it posits that children with ADHD have these skills, but are perhaps unaware of the flexibility and control they have over them. This treatment aims to increase this awareness and subsequently improve ratings of attention, behaviour and other areas of executive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Children with a formal diagnosis of ADHD as given by a psychiatrist or community paediatrician
* Children between the ages of 7 and 11. This age group was selected as previous research on attention training in this population has used this age group
* Children who are currently on a waiting list at a Child and Adolescent Mental Health Service (CAMHS) or a child psychology service, or being seen by a CAMHS or psychology service for medication review only
* Children who speak fluent English which will ensure they are able to comprehend the tasks instructions adequately.

Exclusion Criteria:

* Children who are not stabilised on stimulant medication and/or willing to maintain their medication type/dose
* Children with a major neurological illness or acquired central nervous system injury
* Children who at the point of referral have a co-existing diagnosis of an Autistic Spectrum Disorder
* Children who are currently in receipt of another non-pharmacological intervention for ADHD or who are currently taking part in another research trial

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Inattention on the Swanson, Nolan and Pelham questionnaire (Snap-IV) | Change from baseline in attention post treatment and at follow up 6 weeks later
  Parent's rating of their child's inattentiveness

SECONDARY OUTCOMES:
Hyperactivity on the Swanson, Nolan and Pelham questionnaire (Snap-IV) | Change from baseline in hyperactivity post treatment and at follow up 6 weeks later
  Parent's rating of their child's hyperactivity
Impulsivity on the Swanson, Nolan and Pelham questionnaire (Snap-IV) | Change from baseline in impulsivity post treatment and at follow up 6 weeks later
  Parent's rating of their child's impulsivity
Attentional control on the Attentional Control Scale for Children (ASC-C) | Change from baseline in attentional control post treatment and at follow up 6 weeks later
  Children's self reported ability to focus and shift their attention
Behaviour on the Strengths and Difficulties Questionnaire (SDQ) | Change from baseline in behaviour post treatment and at follow up 6 weeks later
  Parent's ratings of their child's behaviours
Executive functioning on The Behavioural Rating Inventory of Executive Functioning (BRIEF) | Change from baseline in executive functioning post treatment and at follow up 6 weeks later
  Parent's ratings of their child's executive functioning behaviours in the home environment
Working memory on the Weschler Intelligence Scale for Children (WISC-IV) - Digit Span | Change from baseline in working memory post treatment and at follow up 6 weeks later
  Children's Working memory as assessed by the Digit Span subtest
Working memory on the Weschler Intelligence Scale for Children (WISC-IV) - Letter Number Sequencing | Change from baseline in working memory post treatment and at follow up 6 weeks later
  Children's Working memory as assessed by the Letter Number Sequencing subtest
Treatment Acceptability Questionnaire | Rated once at the final session of treatment, 4 weeks after the 2nd baseline is taken
  Parents rating of the acceptability of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wells, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No